CLINICAL TRIAL: NCT05241652
Title: Strong Point of Inspiratory Muscle Training for Kidney and Immune Functions, and Quality of Life of Chronic Kidney Disease Patients on Hemodialysis
Brief Title: Inspiratory Muscle Training for Chronic Kidney Disease Patients on Hemodialysis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitas Padjadjaran (Other)
Responsible Party: Principal Investigator, Irma Ruslina Defi, Principal Investigator, Universitas Padjadjaran
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: IKFR-202201.01
Record Dates: First submitted 2022-01-31; First posted 2022-02-16 (Actual); Last update posted 2023-03-22 (Actual); Status verified 2023-03

CONDITIONS: Chronic Kidney Disease Stage 5 on Dialysis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Active Comparator): Sixteen patients are assigned an IMT exercise program that included inspiratory muscle strengthening exercises thrice a week at a 50% MIP intensity, five sets per time, ten breathing repetitions per set, for an estimated duration of 20 minutes each using Threshold IMT for 12 weeks.
  Interventions: Other: Inspiratory Muscle Training with an intensity of 50% MIP
- Control group (Placebo Comparator): Sixteen patients are assigned an IMT exercise program that included inspiratory muscle strengthening exercises thrice a week at a 10% MIP intensity, five sets per time, ten breathing repetitions per set, for an estimated duration of 20 minutes each using Threshold IMT for 12 weeks.
  Interventions: Other: Inspiratory Muscle Training with an intensity of 10% MIP

INTERVENTIONS:
Other: Inspiratory Muscle Training with an intensity of 50% MIP — Patients received IMT exercise program at a 50% MIP intensity for 12 weeks
  Arms: Intervention group
Other: Inspiratory Muscle Training with an intensity of 10% MIP — Patients received IMT exercise program at a 10% MIP intensity for 12 weeks
  Arms: Control group

SUMMARY:
Chronic Kidney Disease (CKD) is a global public health problem with an increasing prevalence and incidence, poor prognosis, and high costs. It is characterized by changes in the kidney structure and functions for more than three months. It is grouped into several stages, including end-stage kidney disease requiring renal replacement therapy (RRT). Hemodialysis (HD) is one of the RRT options other than kidney transplantation. Regular moderate-intensity exercise may improve certain elements of the immune system and have anti-inflammatory benefits. Aerobic exercise, extremity muscle strength exercises, and inspiratory muscle training have been reported to improve kidney function and quality of life in CKD patients receiving hemodialysis three times a week. However, the effect of inspiratory muscle training on kidney and immune function, and quality of life in CKD patients receiving HD twice a week remains unclear.

DETAILED DESCRIPTION:
Exercise causes a variety of immunological responses, including the production of interleukins. There is some evidence that exercise is correlated with a reduction in systemic inflammation. Prolonged exercise and regular exercise decrease baseline IL-6 levels as a pro-inflammatory cytokine. Inspiratory Muscle Training (IMT) exercise program can improve endothelial function and oxidative stress, both of which affect the progression of kidney disease. The IMT exercise program can induce a decrease in sympathoadrenal activation, as well as a decrease in adrenaline and noradrenaline circulation, thereby preventing endothelial and glycocalyx injury. So, the IMT can improve kidney function. Previous study showed IMT reducing urea and creatinine levels in CKD patients receiving HD thrice a week. The IMT also can improve quality of life of CKD patients receiving HD thrice a week.

Hemodialysis remains the primary RRT modality in Indonesia, and practice is strongly influenced by the socioeconomics of the region due to lack of third-party payers. Stretching resources to maximize outcome benefit is critical, and twice-weekly HD sessions are an improved and cost-effective clinical practice. Observational studies of twice-weekly HD in Taiwan and China have shown a possible benefit of the slower decline of renal function and acceptable nutritional status in recent years. However, there are limited data from performing IMT can improve kidney and immune function, and quality of life of CKD patients receiving HD twice a week.

As result of limited data, the investigators is looked forward to answer about the effect of the IMT exercise program on improving inflammatory cytokine IL-6, kidney function, and quality of life in end-stage CKD patients receiving HD twice a week.

ELIGIBILITY:
Inclusion Criteria:

* can perform inspiratory muscle training (IMT) procedures,
* have a MIP (Maximal Inspiratory Pressure) value of less than 70% of the predicted measurement results using the micro respiratory pressure meter (RPM) tool,
* hemoglobin level greater than 8 g/dL,
* ability to understand oral and written instructions,
* cooperative and willing to participate in the research,
* able to do exercises after signing an informed consent form.

Exclusion Criteria:

* patients with obstructive lung disease, pleural effusion, cardiomegaly, heart failure, coronary heart disease, history of pneumothorax, history of thoracic or abdominal surgery in the last six months, disturbances related to eardrum damage
* have received inspiratory and expiratory muscle training in the past six months
* blood pressure >180/110 mmHg or <80/60 mmHg

Ages: 45 Years to 54 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2022-02-20 (Actual); Primary Completion 2022-04-26 (Actual); Study Completion 2022-05-05 (Actual)

PRIMARY OUTCOMES:
Urea levels | 84 days
  Kidney function will measure with urea and creatinine levels. The level of urea will examine before and 12 weeks after IMT program exercise. The examination is conducted by laboratory staff, followed by the enzymatic method. The urea level in miligrams per deciliter (mg/dL).
Creatinine levels | 84 days
  Kidney function will measure with urea and creatinine levels. The level of creatinine will examine before and 12 weeks after IMT program exercise. The examination is conducted by laboratory staff, followed by the enzymatic method. The creatinine level in miligrams per deciliter (mg/dL).
IL-6 level | 84 days
  Immune function will measure with IL-6 level. The level of IL-6 will examine before and 12 weeks after IMT program exercise. The examination is conducted by laboratory staff, followed by the enzymatic method. The IL-6 levels in picograms per mililiter (pg/ml).
Physical component summary (PCS) | 84 days
  Quality of life will assess using the KDQOL-SFTM v1.3 questionnaire.This questionnaire consists of a physical component summary (PCS), mental component summary (MCS), and kidney disease component summary (KDCS). We will perform interview using the KDQOL-SFTM v1.3 questionnaire before and 12 weeks after IMT program exercise. PCS measure in Unit on Scale with range 0 to 100, higher value mean better outcome.
Mental component summary (MCS) | 84 days
  Quality of life will assess using the KDQOL-SFTM v1.3 questionnaire.This questionnaire consists of a physical component summary (PCS), mental component summary (MCS), and kidney disease component summary (KDCS). We will perform interview using the KDQOL-SFTM v1.3 questionnaire before and 12 weeks after IMT program exercise. MCS measure in Unit on Scale with range 0 to 100, higher value mean better outcome.
Kidney disease component summary (KDCS) | 84 days
  Quality of life will assess using the KDQOL-SFTM v1.3 questionnaire.This questionnaire consists of a physical component summary (PCS), mental component summary (MCS), and kidney disease component summary (KDCS). We will perform interview using the KDQOL-SFTM v1.3 questionnaire before and 12 weeks after IMT program exercise. KDCS measure in Unit on Scale with range 0 to 100, higher value mean better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Irma Ruslina Defi, M.D., Ph.D., Principal Investigator — Universitas Padjadjaran
Locations (1):
- Al Ihsan Province Hospital, Bandung, West Java, Indonesia

REFERENCES:
- [Background] GBD Chronic Kidney Disease Collaboration. Global, regional, and national burden of chronic kidney disease, 1990-2017: a systematic analysis for the Global Burden of Disease Study 2017. Lancet. 2020 Feb 29;395(10225):709-733. doi: 10.1016/S0140-6736(20)30045-3. Epub 2020 Feb 13. PMID 32061315
- [Background] National Kidney Foundation. K/DOQI clinical practice guidelines for chronic kidney disease: evaluation, classification, and stratification. Am J Kidney Dis. 2002 Feb;39(2 Suppl 1):S1-266. No abstract available. PMID 11904577
- [Background] Andrassy KM. Comments on 'KDIGO 2012 Clinical Practice Guideline for the Evaluation and Management of Chronic Kidney Disease'. Kidney Int. 2013 Sep;84(3):622-3. doi: 10.1038/ki.2013.243. No abstract available. PMID 23989362
- [Background] Pellizzaro CO, Thome FS, Veronese FV. Effect of peripheral and respiratory muscle training on the functional capacity of hemodialysis patients. Ren Fail. 2013;35(2):189-97. doi: 10.3109/0886022X.2012.745727. Epub 2012 Nov 30. PMID 23199095
- [Background] Fassbinder TR, Winkelmann ER, Schneider J, Wendland J, Oliveira OB. Functional Capacity and Quality of Life in Patients with Chronic Kidney Disease In Pre-Dialytic Treatment and on Hemodialysis--A Cross sectional study. J Bras Nefrol. 2015 Jan-Mar;37(1):47-54. doi: 10.5935/0101-2800.20150008. English, Portuguese. PMID 25923750
- [Background] Figueiredo RR, Castro AA, Napoleone FM, Faray L, de Paula Junior AR, Osorio RA. Respiratory biofeedback accuracy in chronic renal failure patients: a method comparison. Clin Rehabil. 2012 Aug;26(8):724-32. doi: 10.1177/0269215511431088. Epub 2012 Jan 18. PMID 22257505
- [Background] Peres A, Perotto DL, Dorneles GP, Fuhro MI, Monteiro MB. Effects of intradialytic exercise on systemic cytokine in patients with chronic kidney disease. Ren Fail. 2015;37(9):1430-4. doi: 10.3109/0886022X.2015.1074473. Epub 2015 Aug 14. PMID 26288101
- [Background] Viana JL, Kosmadakis GC, Watson EL, Bevington A, Feehally J, Bishop NC, Smith AC. Evidence for anti-inflammatory effects of exercise in CKD. J Am Soc Nephrol. 2014 Sep;25(9):2121-30. doi: 10.1681/ASN.2013070702. Epub 2014 Apr 3. PMID 24700875
- [Background] Figueiredo PHS, Lima MMO, Costa HS, Martins JB, Flecha OD, Goncalves PF, Alves FL, Rodrigues VGB, Maciel EHB, Mendonca VA, Lacerda ACR, Vieira ELM, Teixeira AL, de Paula F, Balthazar CH. Effects of the inspiratory muscle training and aerobic training on respiratory and functional parameters, inflammatory biomarkers, redox status and quality of life in hemodialysis patients: A randomized clinical trial. PLoS One. 2018 Jul 26;13(7):e0200727. doi: 10.1371/journal.pone.0200727. eCollection 2018. PMID 30048473
- [Background] Bieber B, Qian J, Anand S, Yan Y, Chen N, Wang M, Wang M, Zuo L, Hou FF, Pisoni RL, Robinson BM, Ramirez SP. Two-times weekly hemodialysis in China: frequency, associated patient and treatment characteristics and Quality of Life in the China Dialysis Outcomes and Practice Patterns study. Nephrol Dial Transplant. 2014 Sep;29(9):1770-7. doi: 10.1093/ndt/gft472. Epub 2013 Dec 8. PMID 24322579
- [Derived] Defi IR, Otafirda MV, Novitri N, Rachmi A. Feasibility of inspiratory muscle training as a rehabilitation program for chronic kidney disease patients in a developing country. Eur Rev Med Pharmacol Sci. 2023 Sep;27(18):8330-8339. doi: 10.26355/eurrev_202309_33755. PMID 37782150

DOCUMENTS (2):
  • Study Protocol (2022-05-01): https://cdn.clinicaltrials.gov/large-docs/52/NCT05241652/Prot_000.pdf
  • Statistical Analysis Plan (2022-05-01): https://cdn.clinicaltrials.gov/large-docs/52/NCT05241652/SAP_001.pdf